CLINICAL TRIAL: NCT00860626
Title: Early Response to Interferon Combined Short-Term Nucleoside Analogue Therapy in HBeAg(+) Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: The Third Affliated Hospital of Sun Yat-sen University, The Third Affliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: interferonshorttermnucleoside
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): At the twelfth week of interferon α treatment, HBV DNA is detectable(>1000 copies/ml), or HBeAg is still positive. And nucleoside analogue is added for 12 weeks.
  Interventions: Drug: interferon α plus nucleoside analogue
- 2 (Active Comparator): At the twelfth week of interferon α treatment, HBV DNA is detectable (>1000 copies/ml), or HBeAg is still positive. But no nucleoside analogue is added.
  Interventions: Drug: interferon α
- 3 (Active Comparator): At the twelfth week of interferon α treatment, HBV DNA is undetectable (<1000 copies/ml), or HBeAg is negative. And interferon is continued for another 9 months.
  Interventions: Drug: interferon α

INTERVENTIONS:
Drug: interferon α plus nucleoside analogue — Standard dose of interferon is used for 12 weeks. On 12th week of treatment, HBV DNA is still detectable (>1000 copies/ml), or HBeAg is still positive. And lamivudine is added for 3 months. After nucleoside analogue is added for 3 months, HBV DNA is tested again. If negative, stop nucleoside analogue and use interferon alone for another 6 months or longer. If HBV DNA is still positive, change to another nucleoside analogue or add another nucleoside analogue.
  Arms: 1
Drug: interferon α — Standard dose of interferon is used for 12 weeks.On 12th week of treatment, HBV DNA is still detectable (>1000 copies/ml), or HBeAg is still positive. But no nucleoside analogue is added.
  Arms: 2
Drug: interferon α — Standard dose of interferon is used for 12 weeks.On 12th week of treatment, HBV DNA is undetectable, or HBeAg is negative. And interferon is continued alone for another 9 months.
  Arms: 3

SUMMARY:
For HBeAg(+) patients, interferon is used for 12 weeks. On 12th week of treatment, If HBV DNA is undetectable (<1000 copies/ml), interferon is continued alone for one year. If HBV DNA is still positive, nucleoside analogue is added for 3 months. After nucleoside analogue is added for 3 months, HBV DNA is tested again. If negative, stop nucleoside analogue and use interferon alone for another 6 months or longer. If HBV DNA is still positive, change to another nucleoside analogue or add another nucleoside analogue.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg posive for 6 months
* HBeAg positive, and HBeAb negative
* HBV DNA>1.0×E5 copies/ml
* ALT>80 u/L within 3 months

Exclusion Criteria:

* pregnant women
* conbination infection of HCV, HAV, or HEV
* conbination infection of HIV
* any contraindication of interferon α

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion rate | 3-6 months

SECONDARY OUTCOMES:
HBV DNA loss rate | 3-6 months
HBsAg loss rate | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gao zhiliang, Doctor, Study Chair — The Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China